CLINICAL TRIAL: NCT04269213
Title: A Phase II Study of CPX-351 in Younger Patients < 60 Years Old With Secondary Acute Myeloid Leukemia
Brief Title: CPX-351 for the Treatment of Secondary Acute Myeloid Leukemia in Patients Younger Than 60 Years Old
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 501719; NCI-2019-08946 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 501719 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Acute Myeloid Leukemia With Myelodysplasia-Related Changes; Secondary Acute Myeloid Leukemia; Therapy-Related Acute Myeloid Leukemia
MeSH Terms: interventions — CPX-351; Injections; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (CPX-351) (Experimental): INDUCTION: Patients receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1, 3, and 5 in the absence of disease progression or unacceptable toxicity.
  RE-INDUCTION: Patients who do not achieve remission receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3 in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Beginning 5-8 weeks after the start of the last induction, patients who achieve CR receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3. Treatment repeats every 45 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Liposome-encapsulated Daunorubicin-Cytarabine

INTERVENTIONS:
Drug: Liposome-encapsulated Daunorubicin-Cytarabine — Given IV
  Other Names: CPX-351; Cytarabine-Daunorubicin Liposome for Injection; Liposomal AraC-Daunorubicin CPX-351; Liposomal Cytarabine-Daunorubicin; Liposome-encapsulated Combination of Daunorubicin and Cytarabine; Vyxeos

SUMMARY:
This phase II trial studies how well liposome-encapsulated daunorubicin-cytarabine (CPX-351) works in treating patients with secondary acute myeloid leukemia who are younger than 60 years old. Drugs used in chemotherapy, such as CPX-351, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the complete response rate including morphologic complete remission (CR) and morphologic complete remission with incomplete blood count recovery (CRi) as defined by the International Working Group Criteria.

SECONDARY OBJECTIVE:

I. To determine CR + CRi duration, event free survival (EFS), overall survival (OS), patients successfully proceeding to allogenic hematopoietic cell transplant, and adverse events (AE).

OUTLINE:

INDUCTION: Patients receive liposome-encapsulated daunorubicin-cytarabine intravenously (IV) over 90 minutes on days 1, 3, and 5 in the absence of disease progression or unacceptable toxicity.

RE-INDUCTION: Patients who do not achieve remission receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3 in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Beginning 5-8 weeks after the start of the last induction, patients who achieve CR receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3. Treatment repeats every 45 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, and then every 3 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed:

  * Therapy-related acute myeloid leukemia (AML)
  * AML with antecedent myelodysplastic syndrome (MDS) or chronic myelomonocytic leukemia (CMML)
  * AML with MDS-related changes (as per World Health Organization [WHO])
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Plasma creatinine =< 1.5 x upper limit of normal (ULN)
* Total bilirubin < 2.0 mg/dL
* Serum alanine aminotransferase and aspartate aminotransferase < 3 x ULN
* Left ventricular ejection fraction by echocardiogram or multiple-gated acquisition >= 50%
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Women of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to enrollment and commit to two forms of birth control
* Men must use a latex condom during any sexual contact with women of childbearing potential
* Willing to adhere to protocol specific requirements
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Prior treatment of AML
* Known clinically active central nervous system (CNS) leukemia
* Core-binding factor leukemia
* Acute promyelocytic leukemia
* Uncontrolled other malignancy
* Prior anthracycline exposure > 368 mg/m^2 of daunorubicin or equivalent
* Cardiovascular disease resulting in heart failure (New York Heart Association class III or IV), unstable angina (angina symptoms at rest), or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months
* Hypersensitivity to cytarabine, daunorubicin, or liposomal drugs
* Known active HIV infection
* Known history of active hepatitis B or C infection
* Pre-existing liver disease (e.g. cirrhosis, chronic hepatitis B or C, nonalcoholic steatohepatitis, sclerosing cholangitis)
* Evidence of ongoing, uncontrolled systemic infection
* Pregnant or breastfeeding women
* Subject with concurrent severe and/or uncontrolled medical or psychiatric conditions that in the opinion of the investigator may impair the participation in the study or the evaluation of safety and/or efficacy
* History of Wilson disease or other copper-handling disorders
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2027-01-29 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (morphological complete remission [CR] and incomplete blood count recovery [CRi]) | At day 45
  Defined by the International Working Group Criteria. Will be summarized using frequencies and relative frequencies.

SECONDARY OUTCOMES:
CR + CRi duration | Time from CR or CRi until relapse or last follow-up, assessed up to 5 years
  Will be summarized using standard Kaplan-Meier methods, where estimates of the median obtained with 90% confidence intervals.
Event free survival | Time from treating until disease progression/relapse, death due to disease, or last follow-up, assessed up to 5 years
  Will be summarized using standard Kaplan-Meier methods, where estimates of the median obtained with 90% confidence intervals.
Overall survival | Time from treatment until death due to any cause or last follow-up, assessed up to 5 years
  Will be summarized using standard Kaplan-Meier methods, where estimates of the median obtained with 90% confidence intervals.
Allogeneic hematopoietic cell transplant rate | Up to 5 years
  Transplant rate estimated using a 90% confidence interval obtained using Jeffrey's prior method.
Incidence of adverse events | Up to 5 years
  Will be reported by grade using frequencies and relative frequencies.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Green, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (4):
- United States (4):
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - SUNY Upstate Medical Center, Syracuse, New York
  - Allegheny Health Network Cancer Institute - West Penn Hospital, Pittsburgh, Pennsylvania